CLINICAL TRIAL: NCT03755219
Title: Mesh and Mesh Fixation in Laparoscopic Groin Hernia Surgery: A Swedish Hernia Registry Study
Brief Title: Mesh and Mesh Fixation in Laparoscopic Groin Hernia Surgery
Status: Completed | Type: Observational
Sponsor: Bengt Novik (Other)
Collaborators: Uppsala University (Other); Swedish Hernia Registry (Unknown); Skaraborg Hospital Research & Development Center, Sweden (Unknown)
Responsible Party: Sponsor-Investigator, Bengt Novik, Principal Investigator, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Other Study IDs: Bengan III
Record Dates: First submitted 2018-11-21; First posted 2018-11-27 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Hernia, Inguinal; Surgical Mesh; Laparoscopy; Hernia; Hernia, Femoral; Surgical Procedures, Minimally Invasive; Surgical Staplers; Recurrence; Fixation Device; Complications
Keywords: Totally extraperitoneal; Transabdominal preperitoneal; Fibrin glue; Fibrin sealant; Mesh fixation; Fixation devices
MeSH Terms: conditions — Hernia, Inguinal; Hernia; Hernia, Femoral; Recurrence | interventions — tetraethylpyrazine; tetra-4-amidinophenoxypropane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (8):
- StdPPM: Standard pure polypropylene mesh.
  "Standard" is defined in SHR by weight ≥ 50 g/square meter.
  Interventions: Procedure: TEP; Procedure: TAPP
- LWM: Lightweight mesh: Either a pure polypropylene mesh, or a polypropylene-based composite mesh.
  The study uses SHR's classification of "light-weight" = <50 g/square meter.
  Interventions: Procedure: TEP; Procedure: TAPP
- Tacks, metal: Metal staples or tacks. Material specification of staples/tacks was introduced in SHR 2012.
  Interventions: Procedure: TEP; Procedure: TAPP
- Tacks, absorbable: Absorbable synthetic staples or tacks. Material specification of staples/tacks was introduced in SHR 2012.
  Interventions: Procedure: TEP; Procedure: TAPP
- Tacks, uncategorized: Staples or tacks were in SHR 2005-2011 not further categorized.
  This category also includes staples/tacks registered from 2012 and forth, not being specified as either metal or absorbable.
  Interventions: Procedure: TEP; Procedure: TAPP
- Fibrin glue: Biologic glue/sealant produced from human donor blood
  Interventions: Procedure: TEP; Procedure: TAPP
- Non-fixation: Mesh is deployed without fixation
  Interventions: Procedure: TEP; Procedure: TAPP
- 3D Mesh: Mesh categorized by anatomical shaped, rather than material or weight. Therefore, this category will be excluded in the original study. Depending on the volume of casess found, the 3D mesh category may eventually be analyzed separately in another study..
  Interventions: Procedure: TEP; Procedure: TAPP

INTERVENTIONS:
Procedure: TEP — By laparoscopic (keyhole) approach, the hernia is repaired with a plastic mesh which the surgeon may or may not anchor with some sort of fixation device
  Other Names: Laparoscopic totally extraperitoneal mesh repair
Procedure: TAPP — By laparoscopic (keyhole) approach, the hernia is repaired with a plastic mesh which the surgeon may or may not anchor with some sort of fixation device
  Other Names: Laparoscopic transabdominal preperitoneal mesh repair

SUMMARY:
The study attempts to quantify the relative risks for recurrence depending on complex combinations of plausible risk factors, in particular mesh, mesh fixation, hernia size and hernia type.

For this purpose the investigators will analyze data from the Swedish Hernia Registry (SHR).

DETAILED DESCRIPTION:
This is an open cohort study design where the investigators will analyze existing data that have been prospectively collected in the Swedish Hernia Registry (SHR), which covers > 95% of all groin hernia repairs in Sweden. The very large cohort of more than 38,000 TEP (totally extraperitoneal) and TAPP (transabdominal preperitoneal) repairs enables assessment of the relative risks for recurrence depending on complex combinations of plausible risk factors, in particular mesh, mesh fixation, hernia size and hernia type, with fulfilling statistical power.

Each participant was entered at the date of surgery, when demographic and intraoperative data were registered. Reoperations were registered in the SHR in the same manner as index repairs, and were used as endpoints.

ELIGIBILITY:
Inclusion Criteria:

* All laparoscopic (mainly TEP and TAPP) repairs that have been registered in the SHR from January 1, 2005 until December 31, 2018.

Exclusion Criteria:

* Open repairs.
* Hernioplasties that were converted from laparoscopic to open surgery.
* Age < 15 years.
* Patients not having a 10-digit state-assigned Patient Identification Number.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of all laparoscopic TEP and TAPP repairs that have been registered in the SHR from September 1, 2005 until December 31, 2017.
  The database is the SHR, which was launched in 1992 and prospectively records groin (lateral, medial and femoral) hernia repairs, including both public and private hospitals.
  The source population are all residents in Sweden from the age of 15 years, having a state-assigned personal identity number.
Sampling Method: Non-Probability Sample
Enrollment: 38450 (Actual)
Dates: Start 2005-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Reoperation for recurrence | Assessment at Dec 31, 2018
  The date of the recurrent surgery
Death | Assessment at Dec 31, 2018
  The date of death

CONTACTS AND LOCATIONS:
Overall Officials: Bengt Novik, Principal Investigator — Dept of Clinical Sciences, Karolinska Institutet, Danderyd Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Novik B, Nordin P, Skullman S, Dalenback J, Enochsson L. More recurrences after hernia mesh fixation with short-term absorbable sutures: A registry study of 82 015 Lichtenstein repairs. Arch Surg. 2011 Jan;146(1):12-7. doi: 10.1001/archsurg.2010.302. PMID 21242440
- [Background] Novik B, Hagedorn S, Mork UB, Dahlin K, Skullman S, Dalenback J. Fibrin glue for securing the mesh in laparoscopic totally extraperitoneal inguinal hernia repair: a study with a 40-month prospective follow-up period. Surg Endosc. 2006 Mar;20(3):462-7. doi: 10.1007/s00464-005-0391-3. Epub 2006 Jan 19. PMID 16424986
- [Result] Novik B, et al. Mesh and mesh fixation in laparoscopic groin hernia repairs. A study of 25,189 TEP and TAPP in the Swedish Hernia Registry [congress abstract]. Hernia 2019; 23 (Suppl 2):S251-S252. https://doi.org/10.1007/s10029-019-02013-8
- [Result] Novik B, Sandblom G, Ansorge C, Thorell A. Association of Mesh and Fixation Options with Reoperation Risk after Laparoscopic Groin Hernia Surgery: A Swedish Hernia Registry Study of 25,190 Totally Extraperitoneal and Transabdominal Preperitoneal Repairs. J Am Coll Surg. 2022 Mar 1;234(3):311-325. doi: 10.1097/XCS.0000000000000060. PMID 35213495